CLINICAL TRIAL: NCT05763966
Title: Uppsala Psychosis Cohort: a Multimodal Study in Early Stage Psychosis Patients, High Risk Individuals and Healthy Controls
Brief Title: Uppsala Psychosis Cohort
Acronym: UPC
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UPC_v 1.0
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Early stage psychosis patients (EPP): Diagnosis of psychotic disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) with onset of less than 3 years prior to inclusion.
  Interventions: Other: No intervention
- Individuals at clinical high risk for psychosis (CHR-P): Fulfills criteria for clinical high risk for psychosis according to Structured Interview for Psychosis-risk Syndromes (SIPS).
  Interventions: Other: No intervention
- Healthy controls (HC): Age- and sexmatched controls.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study where participants are followed over time

SUMMARY:
A multimodal longitudinal study in early stage psychosis patients and individuals at high risk for psychosis. Healthy controls are included for baseline comparisons. The aim is to investigate disease mechanisms of psychotic disorders, specifically focusing on the synaptic pruning hypothesis.

DETAILED DESCRIPTION:
This is a single-site observational study examining synaptic density using positron emission tomography (PET) and the radioligand [18F]SynVest-1 binding to the synaptic vesicle glycoprotein 2A. In addition to PET, the study includes clinical assessment, cognitive testing, multimodal magnetic resonance imaging (MRI) measures, neurophysiological measures, lumbar punction for cerebrospinal fluid (CSF) analyses, blood sampling, heart rate variability measures. Early stage psychosis patients and clinical high-risk individuals are subject to repeat assessment after 1 year (including PET), and at 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria

For EPP:

* Diagnosis as assessed using DSM-5 of one of the following: schizophrenia, schizophreniform psychosis, psychosis not otherwise specified (NOS), brief psychosis, schizoaffective syndrome, delusional disorder
* Onset of psychotic symptoms together with functional decline no more than 3 years prior to inclusion visit

For CHR-P:

Clinical high risk for psychosis as determined using Structured Interview for Psychosis-risk Syndromes (SIPS).

Exclusion Criteria

For EPP and CHR-P:

* Other dominant psychiatric illness that is deemed to be related to current psychotic symptoms (including bipolar disorder, major depressive disorder, autism)
* Long-term daily treatment (<2 weeks) with benzodiazepines, such that there is an inability to refrain from treatment during testing procedures.

For HC:

* A history of diagnosis of a major psychiatric disorder, including substance use disorders.
* A family history of psychotic disorders or bipolar disorder in first degree relatives.

For all participants:

* Evidence based on medical history, clinical signs, MRI or laboratory tests of clinically significant somatic disorder, or previous disorder with brain engagement (e.g. tumour, neuroinflammatory disease, epilepsy) or significant brain trauma.
* Exposure to an effective radiation dose of 25 mSv during the past year.
* Pregnancy, lactating or breastfeeding (women).
* Lack of proficiency in Swedish language, or documented intellectual disability that prohibits ability to give informed consent.
* Meets diagnostic criteria of substance use disorder (excluding nicotine dependence) as assessed using DSM-5 or as determined using repeated positive urine screens during the course of the study.
* Metallic object in the eye, or ferro/electromagnetic implants. History of claustrophobic anxiety during MRI.
* Symptoms of severe bacterial, fungal, or viral infection (including upper respiratory tract infection), with systemic effects as detected by e.g. fever, within 7 days prior to inclusion.
* Treatment with any antihemostatic medication within 2 weeks of lumbar puncture and arterial line placement of either the baseline or 1 year follow-up.
* Blood donation (1 unit or more) within 90 days prior to Screening, plasma donation from 1 week prior to Screening, and platelet donation from 6 weeks prior to inclusion.
* Other unspecified reasons that, in the opinion of the Investigator or the Sponsor, make the participant unsuitable for enrollment. This may include very high symptom severity or signs of aggressiveness and hostility.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Early stage Psychosis Patients (EPP) (<3 year duration) and individuals at clinical high risk for psychosis (CHR-P) are recruited from the psychiatry clinic. Healthy controls (HC) are recruited by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Synaptic density in early stage psychosis (EPP) patients and individuals at Clinical High Risk for Psychosis (CHR-P) compared to healthy controls (HC). | 1 timepoint (baseline)
  Group comparisons of [18F]SynVesT-1 binding to the synaptic vesicle glycoprotein 2A (SV2A) at baseline between EPP, CHR-P and HC.
Changes in synaptic density in EPP and CHR-P between baseline and after 1 year. | 1 year
  Comparison of regional [18F]SynVesT-1 binding to SV2A between baseline and follow-up in EPP and CHR-P.
Measures of cognitive function, magnetic resonance imaging (MRI), electroencephalogram (EEG) in relation to SV2A in EPP, CHR-P and HC. | 1 timepoint (baseline)
  Analyses of group differences and correlational analyses between cognitive performance as measured using Measurement and Treatment Research to Improve Cognition in Schizophrenia battery (MATRICS), MRI measures of connectivity and metabolite levels, and EEG measures of cortical excitability to [18F]SynVesT-1 binding to SV2A will be performed in EPP, CHR-P and HC.
Measures of cognitive function, magnetic resonance imaging (MRI), electroencephalogram (EEG) in relation to changes in SV2A in EPP and CHR-P. | 1 year
  Analyses of group differences and correlational analyses between cognitive performance as measured using MATRICS, MRI measures of connectivity and metabolite levels, and EEG measures of cortical excitability to longitudinal differences in [18F]SynVesT-1 binding to SV2A will be performed in EPP and CHR-P.
Candidate disease markers in cerebrospinal fluid in relation to SV2A in EPP, CHR-P and HC. | 1 timepoint (baseline)
  Analyses of group differences and correlational analyses between candidate disease markers in CSF to [18F]SynVesT-1 binding to SV2A will be performed in EPP, CHR-P and HC.
Candidate disease markers in cerebrospinal fluid in relation to changes in SV2A in EPP and CHR-P. | 1 year
  Analyses of group differences and correlational analyses between candidate disease markers in CSF to changes in [18F]SynVesT-1 binding to longitudinal differences in [18F]SynVesT-1 binding to SV2A will be performed in EPP and CHR-P.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Cervenka, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available to other researchers upon request, as allowed by national legislation.